CLINICAL TRIAL: NCT05993312
Title: Quality of Life in Traumatic Brain Injury Patients: Assessment at Discharge From an Intensive Care Unit.
Brief Title: Quality of Life in Traumatic Brain Injury Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Principal Investigator, Hedi Gharsallah, DR Aicha REBAI, General Administration of Military Health, Tunisia
Other Study IDs: QLTBIP
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: All Adult Patients Admitted to theHMPIT ICU for Management of Head Trauma
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A bras actif
  Interventions: Other: quality of life

INTERVENTIONS:
Other: quality of life — To describe the relationship between distant sequelae of trauma assessed by the GOSE scale and quality of life

SUMMARY:
The aim of this study is to describe the quality of life of CT patients in our study, at least 6 months after the occurrence of the trauma. This assessment is related to the patient's degree of sequelae, using the GOSE scale.

DETAILED DESCRIPTION:
The assessment of patients quality of life would appear to be a particularly relevant tool in the ongoing drive to improve the quality of care. Thus, we should no longer simply assess how patients "should feel", based on objective biomedical criteria, but how they actually "perceive" themselves, based on subjective criteria.

This is particularly true in the case of traumatic brain injury , which is a high-incidence pathology with significant morbidity and mortality consequences that can lead to permanent sequelae . While research over the past 30 years has focused on the neuropsychological and functional outcomes of this event, less is known about the views of head injury survivors and their families on their quality of life, subjective well-being and related factors.

The aim of this study is to describe the quality of life of CT patients at least 6 months after the trauma. This assessment is related to the patient's degree of sequelae, using the Glasgow Outcome Scale Extended GOSE.

ELIGIBILITY:
Inclusion Criteria:

All adult patients (age 18 or over) admitted to the HMPIT intensive care unit for management of head trauma (isolated or as part of a polytrauma).

Exclusion Criteria:

Patients lost to follow-up after discharge. Incomplete ICU medical records. Patients or their families who refused to participate in the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Collection of patients: medical data from the ICU medical record. Data collection of quality of life : outpatient clinic: the interview will be conducted by telephone.
  If number phone patient cannot be reached, the questionnaire will be sent by post to the patient's address
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
quality of life in patients with BI / The short form12 SF12 questionnaire | 6 month
  To describe the relationship between distant sequelae of trauma assessed by the GOSE scale and quality of life in patients with BI.

CONTACTS AND LOCATIONS:
Overall Officials: Aicha N REBAI, Study Chair — hopital militaire de TUNIS
Locations (2):
- Tunisia (2):
  - Military Hospital of Tunis, Tunis, Montfleury
  - Service de réanimation, Tunis, Montfleury

IPD SHARING:
Plan to Share IPD: Undecided